CLINICAL TRIAL: NCT00006330
Title: Pharmacokinetic and Pharmacodynamic Interaction Study of Digoxin and Hawthorn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCRR-M01RR00042-1693; M01RR000042 (NIH)
Record Dates: First submitted 2000-10-04; First posted 2000-10-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-11

CONDITIONS: Heart Diseases
Keywords: Digoxin; Effect modifiers (Epidemiology); Rosales; Drug Interaction
MeSH Terms: conditions — Heart Diseases | interventions — Digoxin; crataegus extract

INTERVENTIONS:
Drug: Digoxin
Drug: Hawthorn

SUMMARY:
Hawthorn (Crataegus oxyacantha) is a natural product that is popular in European and American herbal medicine practice. Some of its cardiac uses include the treatment of high and low blood pressure, rapid heart beat, chest pain, and blocked arteries. In many cases, it is used as an adjuvant agent with other cardiac drugs such as digoxin, amiodarone, and warfarin. To date, little information is known about the effect of hawthorn when taken with other drugs and if toxicities occur when hawthorn is used with other drugs. The purpose of this study is to examine the interaction between digoxin and hawthorn in eight healthy subjects. Subjects will be recruited by advertisement. The design of the study will include a 10-day and a three-week treatment phase of digoxin 0.125 mg - 0.25 mg/day and hawthorn (Crataegus special extract WS1442, Schwabe Co.) 450 mg twice daily or placebo, with a randomized crossover. There will be a three-week washout period in between treatment phases. On day 10 (phase I) and day 21 (phase II), subjects will have 12 blood samples drawn for pharmacokinetic analysis. The plasma samples will be measured for digoxin concentration. Additionally, the subjects will be assessed for any clinical toxicities or adverse events. The significance of this study is to provide the clinician with information regarding the safe use of digoxin in combination with the herbal supplement, hawthorn.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult
* Not regularly taking any prescription or non-prescription medications (including natural products or supplements) and is willing to avoid all medications other than the study drugs during the study period.
* Willing to avoid drinking any alcohol throughout the study period.
* Does not currently smoke and is willing to avoid smoking during the study period.
* Willing to adhere to dietary restrictions as required during the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Univ. of Michigan Medical Center, Ann Arbor, Michigan, United States